CLINICAL TRIAL: NCT06169917
Title: Potential Influences of Respiration Patterns on Experimental Pain Sensitization
Brief Title: Pain Processing In Relation To Breathing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Schweinhardt Petra, Prof. Dr. med, Balgrist University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-00518
Record Dates: First submitted 2023-09-04; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Central Sensitisation; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy participants (Experimental): Participants should be aged 18-40, in good health, capable of informed consent, without major medical/psychiatric conditions (e.g., heart disease, diabetes, autoimmune disorders, infectious diseases, major depressive disorder), chronic pain, respiratory issues, or ongoing acute pain, qualify. Exclusions: inability to follow instructions (e.g., language issues), recent alcohol/drug/analgesic use (<24h), caffeine intake (>100mg <8h), or scar tissue/general reduced sensitivity in test areas.
  Participants undergo three interventions. The heat stimulation intervention is performed twice. During one heat stimulation intervention, participants receive the 'resonance frequency breathing' intervention. During the other heat stimulation intervention, participants receive the 'natural frequency breathing' intervention. The order of the breathing interventions is counterbalanced across participants.
  Interventions: Behavioral: Paced Resonance Frequency Breathing; Behavioral: Paced Breathing at Natural Frequency; Other: Heat Stimulations

INTERVENTIONS:
Behavioral: Paced Resonance Frequency Breathing — Participants are required to pace their breathing to their pre-determined individual resonance frequency.
Behavioral: Paced Breathing at Natural Frequency — Participants are required to pace their breathing to their pre-determined individual breathing frequency at rest.
Other: Heat Stimulations — Participants will undergo a heat stimulation procedure on their left and right foot (the order of which is counterbalanced across participants). During this procedure, there are 10 blocks, with an inter-stimulus interval of 30 seconds between two blocks. During a block, six 6-second heat stimulations (48 degrees) are given. Between the stimulations, the temperature quickly returns to baseline (32 degrees).

SUMMARY:
The goal of this clinical trial is to investigate the effect of breathing on the processing of experimental pain in healthy participants. The main questions are:

1. Does breathing rate influence the spatial extent of thermally induced secondary hyperalgesia, a proxy of central sensitization?
2. Does resonance frequency breathing influence the autonomic nervous system, compared to baseline and compared to paced breathing at a natural frequency?
3. Is spinal excitability, measured using the magnitude of the nociception withdrawal reflex (NWR), affected by resonance frequency breathing, compared to paced breathing at a natural frequency?

Participants:

* will receive heat stimuli
* 's skin's sensitivity will be tested using quantitative sensory testing tools.
* will receive various instructions on the speed of their breathing
* 's heart rate, respiratory rate and sweat response will be measured
* will fill in questionnaires

Researchers will compare the spatial extent of sensitivity resulting from application of heat stimuli during paced resonance frequency breathing compared to paced breathing at a natural frequency to see if the breathing rhythm influences central sensitization processes.

ELIGIBILITY:
Inclusion Criteria:

1. over 18 and below 40 years of age
2. good general health
3. able to give informed consent

Exclusion Criteria:

1. any major medical or psychiatric condition (e.g. heart disease, diabetes, autoimmune disorders, infectious diseases, major depressive disorder), any chronic pain condition, any respiratory problems, any current acute pain at time of study
2. inability to follow study instructions, e.g. due to language problems
3. Consumption of alcohol, drugs, analgesics within the last 24 h
4. Consumption of no more than 100 mg of caffeine within the last 8 h
5. Scar tissue or generally reduced sensitivity in the designated testing site areas

Additional exclusion criteria for experiments 3 and 4

1. Shoe size < 38
2. Restless-Legs-Syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-14 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Area of Hypersensitivity surrounding the primary stimulation site | 40 minutes
  Before and after thermal stimulations, the sensitivity of the skin is tested using a von Frey Filament, a Pin Prick and a brush. Thermal stimulations cause hypersensitivity of the skin, resulting in an area of hypersensitivity surrounding the stimulation site. The primary outcome measure is the amount of change in the area of hypersensitivity from before to after the thermal stimulations. The measuring unit of this outcome is square centimetres.

SECONDARY OUTCOMES:
Power in the Low-frequency Range of the Heart Rate Variability | 25 minutes
  Power is measured in units of milliseconds squared (ms 2) for a the low frequency band (Hz), ranging from 0.04 - 0.15Hz
Root Mean Square of Successive Differences of the Heart Rate Variability | 25 minutes
  The measuring unit to measure heart rate variability is the root mean square of successive differences between normal heartbeats.
Galvanic Skin Potential | 25 minutes
  Galvanic Skin potential is taken as a reflection of electrodermal activity. The measuring unit of this outcome is microsiemens
Threshold and Magnitude of the Nociceptive Withdrawal Reflex | 25 minutes
  The nociceptive withdrawal reflex is triggered using an supratheshold electrical stimulation at the nervus suralis leading muscle contraction in the ipsilateral biceps femoris, rectus femoris and tibialis anterior. Muscle contraction is measures in millivolt using electromyogram with recording electrodes attached to the respective muscles

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Balgrist, University Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided